CLINICAL TRIAL: NCT04213820
Title: TMS Treatment for Anorexia Nervosa: Effects on Body Image Processing and Clinical Outcome Measures
Brief Title: TMS and Body Image Treatment for Anorexia Nervosa
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Region Östergötland (Other)
Responsible Party: Principal Investigator, Maria Zetterqvist, Principal Investigator, Region Östergötland
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2019-02821
Record Dates: First submitted 2019-12-27; First posted 2019-12-30 (Actual); Last update posted 2023-08-29 (Actual); Status verified 2023-08

CONDITIONS: Anorexia Nervosa
MeSH Terms: conditions — Anorexia Nervosa | interventions — Transcranial Magnetic Stimulation; Therapeutics

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Treatment as usual (Active Comparator): Participants will receive treatment as usual at the eating disorder unit at the Child and adolescent psychiatric clinic and at the Psychiatric clinic during 4 weeks.
  Interventions: Behavioral: Treatment as usual
- TMS and body image intervention (Experimental): Participants will receive TMS and a body image intervention daily 5 times/week during 4 weeks
  Interventions: Device: Transcranial magnetic stimulation; Behavioral: Body Image Intervention
- sham TMS and body image intervention (Sham Comparator): Participants will receive sham TMS and a body image intervention Daily 5 times/week during 4 weeks
  Interventions: Behavioral: Body Image Intervention

INTERVENTIONS:
Device: Transcranial magnetic stimulation — TMS (theta burst) will be administered consisting of bursts containing 3 pulses at 50 Hz and an intensity of 80% motor threshold repeated at 200 ms intervals (i.e., at 5 Hz) and a 10 s between burst triplet interval for a total for 190 s (600 pulses). The intervention will be given daily 5 times/week during 4 weeks.
  Arms: TMS and body image intervention
Behavioral: Body Image Intervention — Body image interventions delivered directly after TMS will include body exercises that target disturbed body image and psychoeducation about the body. Together with a therapist the participants with anorexia nervosa will explore and estimate their body size through feedback.
  Arms: TMS and body image intervention; sham TMS and body image intervention
Behavioral: Treatment as usual — Treatment as usual at the eating disorder unit, Child and adolescent psychiatric clinic and Psychiatric clinic is delivered during 4 weeks
  Arms: Treatment as usual

SUMMARY:
To evaluate if TMS together with a body image intervention is an efficacious treatment for anorexia nervosa compared to treatment as usual.

ELIGIBILITY:
Inclusion Criteria:

* Being enrolled as a patient at the eating disorder unit of the Child and adolescent psychiatric clinic and Psychiatric clinic in Linköping
* Having a DSM-5 diagnosis of anorexia nervosa, atypical anorexia (restrictive type)
* Being at least 18 years of age
* Having a BMI of 20 or under.
* Being free of psychotropic medications or on stable (at least three months on the same dose) medication.

Exclusion Criteria:

* Clinical diagnosis of schizophrenia or psychotic disorder
* Clinical diagnosis of bipolar disorder
* Alcohol/drug dependence
* Ongoing treatment with antipsychotics or tricyclic antidepressants
* Previous severe head injury
* Birth before 33 weeks of gestation
* Hearing impairment
* Earlier epilepsy or seizures of other causes
* Having severe claustrophobia
* Being pregnant
* Having a cognitive disability

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2019-09-25 (Actual); Primary Completion 2024-02 (Estimated); Study Completion 2024-02 (Estimated)

PRIMARY OUTCOMES:
Eating Disorder Examination Questionnaire (EDE-Q) | Change from baseline at 4 weeks and at 6 months
  EDE-Q measures symptoms of eating disorder. It contains at total of 36 items. 23 of these are rated on a Likert scale between 0-6 and contains 4 subscales: Restraint (ranging from 0-30); Eating concern (ranging from 0-30); shape concern (ranging from 0-48); weight concern (ranging from 0-30). Higher scores indicating more difficulties with eating disorder. In addition, 11 open ended questions concern binge eating and compensating behaviors.
Body Attitude Test (BAT) | Change from baseline at 4 weeks and at 6 months
  BAT measures attitudes toward one own body. It contains a total of 20 items that are rated on a Likert scale between 0-5. Total scores range from 0-100. Higher scores indicate more problems with body attitude.
Body Shape Questionnaire (BSQ) | Change from baseline at 4 weeks and at 6 months
  BSQ measures dissatisfaction with one's own body/figure. It contains a total of 34 items, which are rated on a Likert scale ranging from 1-6. total scores range from 34-204, with higher scores indicating more dissatisfaction.
Figure Rating Scale | Change from baseline at 4 weeks and at 6 months
  Figure Rating Scale measures body image and estimation of one's own body size. Each figure presents nine schematic silhouettes, ranging from extreme thinness (1) to extreme obesity (9). For research purposes, participants are asked to self-select the silhouette that best indicates his or her current body size (ranging from 1-9) and the silhouette that reflects his or her ideal body size (ranging from 1-9).
Body Mass Index (BMI) | Change from baseline at 4 weeks and at 6 months
  Body Mass Index is a person's weight in kilograms divided by the square of height in meters and is an indication of under- or overweight in adults.

OTHER OUTCOMES:
Extrastriatal body area (EBA) activation during fMRI | Change from baseline at 4 weeks and at 6 months
Extrastriatal body area (EBA) connectivity during resting state fMRI | Change from baseline at 4 weeks and at 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Maria A Zetterqvist, PhD, Principal Investigator — Region Östergötland/Linköping university
Locations (1):
- Region Östergötland BUP-kliniken, Linköping, Sweden

IPD SHARING:
Plan to Share IPD: No